



## **Participant Consent Form**

Validating neuro-navigated TMS stimulation in chronic SCI patients: a feasibility study towards a gene therapy for SCI.

**IRAS Number: 320531** 

**Chief Investigator: Mr Aminul Ahmed** 

Participant Identification Number for this trial:

| I confirm that I have read the information sheet (version 1 dated 28/02/2023) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from the sponsor of the trial (King's College London/King's College Hospital NHS Trust and responsible persons authorised by the sponsor, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. I agree to my General Practitioner being informed of my participation in the study I agree to be contacted about ethically approved future research. Name of Participant Date Signature Name of Person Date Signature | | | | | Please<br>initial bo |
|---|---|---|---|---|---|
| I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from the sponsor of the trial (King's College London/King's College Hospital NHS Trust and responsible persons authorised by the sponsor, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. I agree to my General Practitioner being informed of my participation in the study I agree to be contacted about ethically approved future research. Name of Participant Date Signature Name of Person Date Signature | 1 | I confirm that I have read the | e information sheet (version | on 1 dated 28/02/2023) for the above study | IIIILIAI DO |
| answered satisfactorily. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from the sponsor of the trial (King's College London/King's College Hospital NHS Trust and responsible persons authorised by the sponsor, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. I agree to my General Practitioner being informed of my participation in the study I agree to be contacted about ethically approved future research. Name of Participant Date Signature Name of Person Date Signature | | | | | |
| I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from the sponsor of the trial (King's College London/King's College Hospital NHS Trust and responsible persons authorised by the sponsor, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. I agree to my General Practitioner being informed of my participation in the study I agree to be contacted about ethically approved future research. Name of Participant Date Signature Name of Person Date Signature | | | | | |
| giving any reason, without my medical care or legal rights being affected. I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from the sponsor of the trial (King's College London/King's College Hospital NHS Trust and responsible persons authorised by the sponsor, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. I agree to my General Practitioner being informed of my participation in the study I agree to be contacted about ethically approved future research. I agree to take part in the above study. Name of Participant Date Signature Name of Person Date Signature | | | | | |
| I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from the sponsor of the trial (King's College London/King's College Hospital NHS Trust and responsible persons authorised by the sponsor, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. I agree to my General Practitioner being informed of my participation in the study I agree to be contacted about ethically approved future research. Name of Participant Date Signature Name of Person Date Signature | | | | | |
| be looked at by individuals from the sponsor of the trial (King's College London/King's College Hospital NHS Trust and responsible persons authorised by the sponsor, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. I agree to my General Practitioner being informed of my participation in the study I agree to be contacted about ethically approved future research. Name of Participant Date Signature Name of Person Date Signature | _ | | | | |
| Hospital NHS Trust and responsible persons authorised by the sponsor, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. I agree to my General Practitioner being informed of my participation in the study I agree to be contacted about ethically approved future research. I agree to take part in the above study. Name of Participant Date Signature Name of Person Date Signature | 3 | | | | |
| or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. I agree to my General Practitioner being informed of my participation in the study I agree to be contacted about ethically approved future research. I agree to take part in the above study. Name of Participant Date Signature Name of Person Date Signature | | be looked at by individuals from the sponsor of the trial (King's College London/King's College | | | |
| these individuals to have access to my records. I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. I agree to my General Practitioner being informed of my participation in the study I agree to be contacted about ethically approved future research. I agree to take part in the above study. Name of Participant Date Signature Name of Person Date Signature | | Hospital NHS Trust and responsible persons authorised by the sponsor, from regulatory authorities | | | |
| I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. I agree to my General Practitioner being informed of my participation in the study I agree to be contacted about ethically approved future research. I agree to take part in the above study. Name of Participant Date Signature Name of Person Date Signature | | or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for | | | |
| future, and may be shared anonymously with other researchers. I agree to my General Practitioner being informed of my participation in the study I agree to be contacted about ethically approved future research. I agree to take part in the above study. Name of Participant Date Signature Name of Person Date Signature | | these individuals to have access to my records. | | | |
| I agree to my General Practitioner being informed of my participation in the study I agree to be contacted about ethically approved future research. I agree to take part in the above study. Name of Participant Date Signature Name of Person Date Signature | 4 | I understand that the information collected about me will be used to support other research in the | | | |
| I agree to be contacted about ethically approved future research. I agree to take part in the above study. Name of Participant Date Signature Name of Person Date Signature | | future, and may be shared anonymously with other researchers. | | | |
| I agree to be contacted about ethically approved future research. I agree to take part in the above study. Name of Participant Date Signature Name of Person Date Signature | 5 | I agree to my General Practitioner being informed of my participation in the study | | | |
| 7 I agree to take part in the above study. Name of Participant Date Signature Name of Person Date Signature | | | | | |
| Name of Participant Date Signature Name of Person Date Signature | 6 | I agree to be contacted about ethically approved future research. | | | |
| Name of Participant Date Signature Name of Person Date Signature | | | | | |
| Name of Person Date Signature | 7 | I agree to take part in the above study. | | | |
| Name of Person Date Signature | | | | | |
| Name of Person Date Signature | | | | | |
| Name of Person Date Signature | | | | | |
| Name of Person Date Signature | | | | | |
| • | | Name of Participant | Date | Signature | |
| • | | | | | |
| • | | | | | |
| taking consent | | Name of Person | Date | Signature | |
| | | taking consent | | | |

When completed: 1 for participant; 1 for researcher site file; 1 (original) to be kept in medical notes.